CLINICAL TRIAL: NCT00130494
Title: Multicenter, Open-label, Randomized Phase III Trial for Administration of Zoledronate to Breast Cancer Metastatic Patients With Non-symptomatic Bone Lesions
Brief Title: Zoledronic Acid Administration to Metastatic Breast Cancer Patients With Non-symptomatic Bone Lesions
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM 2001-05
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer; Neoplasm Metastasis
Keywords: Non-symptomatic bone metastases.
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Zoledronic Acid

ARMS (2):
- Arm A: Zoledronic acid 4 mg (Experimental): Zoledronate 4 mg every 3 or 4 weeks. This arm will receive study treatment from the time of entry into the trial, until the appearance of the symptoms of bone metastases (or a maximum period of 12 months, whichever occurs first).
  Interventions: Drug: Zoledronic acid
- Arm B: Observation (No Intervention): Patients will not receive any treatment with bisphosphonates until the time of onset of symptoms (or a maximum period of 12 months, whichever occurs sooner).

INTERVENTIONS:
Drug: Zoledronic acid
  Other Names: Zometa
  Arms: Arm A: Zoledronic acid 4 mg

SUMMARY:
This is an open-label, randomized, multicenter phase III trial to assess the efficacy of early administration of zoledronate versus observation in delaying bone-related symptoms in metastatic breast cancer patients.

DETAILED DESCRIPTION:
Patients will be randomised to receive 4 mg zoledronate every 3-4 weeks versus observation until bone-related symptoms appear, or up to 12 months. One hundred twelve patients per treatment arm will be enrolled in the study.

Once bone-related symptoms appear, study participation is over. During the study, the following will be assessed:

* quality of life,
* performance status,
* pain rating,
* analgesic administration and
* adverse events The principal objective is the delay in bone-related symptoms in those patients with early zoledronate administration.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Age >= 18 years old.
* Metastatic breast cancer patients with lytic, sclerotic or mixed bone lesions.
* Non-symptomatic bone lesions, defined as pain absence, lack of bone complications (fracture, hypercalcemia, Central Nervous System (CNS) compression), no need of analgesic chronic administration for bone disease.
* A maximum of two chemotherapy lines for metastatic disease.
* A maximum of two hormone therapy lines for metastatic disease.
* Normal, minimally altered renal function (serum creatinine < 1.5 x Upper Normal Limit (UNL)).
* Normal serum calcium levels.
* Performance status 0,1 (World Health Organization (WHO)).
* Negative pregnancy test before study recruitment.

Exclusion Criteria:

* Previous treatment with bisphosphonates or raloxifene in the 30 days prior to randomization.
* Metastasis in CNS.
* History of hypersensitivity to bisphosphonates.
* Pregnant or lactating women.
* Third chemotherapy line for metastatic disease.
* Third hormone therapy line for metastatic disease.
* Males.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2002-08-29 (Actual); Primary Completion 2006-11-20 (Actual); Study Completion 2007-10-22 (Actual)

PRIMARY OUTCOMES:
Time to first bone metastases | Up to disease progression
  The main variable of evaluation is the time until the appearance of first bone metastases.

SECONDARY OUTCOMES:
Quality of life per treatment arm | Up to disease progression
  Quality of Life (QoL) will be measured with Short Form (SF)-36 questionnaire and Short questionnaire for the evaluation of pain since baseline visit and during all treatment period delivered to the patient before the start of each visit.
The Number of Participants Who Experienced Adverse Events (AE) | Through study treatment
  Safety will be assessed by standard clinical and laboratory tests. Adverse events grade will be defined by the NCI CTCAE.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital Clínico Universitario de Valencia; Study Director, Study Director — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Spanish Breast Cancer Research Group (GEICAM), San Sebastián de los Reyes, Madrid, Spain

REFERENCES:
- See also: Click here for more information about this study: GEICAM 2001-05 — http://www.geicam.org